CLINICAL TRIAL: NCT04026581
Title: Real World Testing of a Brain-Computer Interface to Operate a Commercial Augmentative and Alternative Communication System
Brief Title: Real World Testing of a Brain-Computer Interface
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Katya Hill, Associate Professor, University of Pittsburgh
Other Study IDs: STUDY19010094; 90IFDV0002-01-00 (Other Grant/Funding Number: NIDILRR)
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Amyotrophic Lateral Sclerosis; Brain Stem Stroke; Cerebral Palsy; Traumatic Brain Injury; Speech Disorders
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Brain Stem Infarctions; Cerebral Palsy; Brain Injuries, Traumatic; Speech Disorders | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Assessment: A comprehensive AAC assessment collecting clinical and personal data required to select a speech-generating device (SGD) is conducted along with a trial of three AAC technology solutions, followed by a trial for BCI access to an AAC system.
  Interventions: Behavioral: Speech generating device (SGD) evaluation including BCI access
- Training and Treatment: AAC training and treatment services will be provided and communication performance outcomes monitored over the course of studying clinical treatment services. At monthly home visits the SLP gathers clinical and personal data on communication performance outcomes and user satisfaction of their AAC system and any alternative access methods.
  Interventions: Behavioral: Training and treatment

INTERVENTIONS:
Behavioral: Speech generating device (SGD) evaluation including BCI access — At the initial evaluation the participants will review the full range of AAC options and speech generating devices (SGDs) and complete a speech and language evaluation. The second evaluation date will involve a trial of SGDs matched to the participant's assessment results. The third visit is the trial of an AAC system with BCI access. Should the dry electrode headgear for BCI access prove ineffective, then the gel electrode cap will be offered to the participant for trial. At the end of the third visit, the evaluation results will be discussed with participant and family, and they will be asked to select the preferred SGD.
  Groups: Assessment
Behavioral: Training and treatment — Participants receive training on the selected SGD followed by monthly treatment sessions from the SLP who monitors performance. In some cases the participants' SGD will be an AAC system with BCI access. In this case training will also include an identified system support person. Use of the SGD is monitored on a monthly basis through home visits and/or tele-practice sessions, when requested. Technical support for the SGD is provided on an as needed basis or when requested by the participant or support person.
  Groups: Training and Treatment

SUMMARY:
The goal of this project is to test a new AAC-BCI device comparing gel and dry electrode headgear used for communication while providing clinical care. Innovative resources will be employed to support the standard of care without considering limitations based on service billing codes. Clinical services will include AAC assessment, AAC-BCI device and treatment to individuals with minimal movement due to amyotrophic lateral sclerosis (ALS), brain stem strokes, severe cerebral palsy, traumatic brain injury (TBI) and their family support person. This is a descriptive study designed to measure and monitor the communication performance of individuals using the AAC-BCI, any other AAC strategies, their user satisfaction and perceptions of communication effectiveness, and the satisfaction of the family support persons.

DETAILED DESCRIPTION:
This clinical trial follows a descriptive study design collecting data to measure and monitor variables related to the standard of care in providing speech language pathology augmentative and alternative communication clinical (AAC) assessment and treatment. The study tracks participants through the AAC, speech generating device trial and AAC-BCI trial processes. In addition this study measures and monitors the communication performance of individuals using the AAC-BCI and any other AAC strategies for treatment in the home. Data on communication performance, user satisfaction, and perceptions of communication effectiveness are gathered over monthly visits along with the satisfaction and perceptions of communication effectiveness by the family support persons.

ELIGIBILITY:
Inclusion Criteria:

* natural speech does not meet daily communication needs requiring using a speech generating device
* Has a diagnosis resulting in minimal movement interfering with direct selection to a keyboard or AAC display
* age 14 and above
* able to read a standard computer screen
* able to follow instructions
* English as their native language

Exclusion Criteria:

* history of photosensitive epilepsy
* open sores on the scalp
* history of uncorrectable hearing loss
* unavailable to participate during the times scheduled for the study

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with severe communication disabilities and minimal movement impairment.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change in daily communication performance | Baseline vs. 1 month
  Monitoring daily use of a speech generating device (SGD) for communication. Average communication rate based on total number of words used during the day.
Change in daily communication performance | 1 month vs. 2 months
  Monitoring daily use of a speech generating device (SGD) for communication. Average communication rate based on total number of words used during the day.
Change in daily communication performance | 2 months vs. 3 months
  Monitoring daily use of a speech generating device (SGD) for communication. Average communication rate based on total number of words used during the day.
Change in daily communication performance | 3 months vs. 4 months
  Monitoring daily use of a speech generating device (SGD) for communication. Average communication rate based on total number of words used during the day.
Change in daily communication performance | 4 months vs. 5 months
  Monitoring daily use of a speech generating device (SGD) for communication. Average communication rate based on total number of words used during the day.
Change in daily communication performance | 5 months vs. 6 months
  Monitoring daily use of a speech generating device (SGD) for communication. Average communication rate based on total number of words used during the day.
Change in daily communication performance | 6 months vs. 7 months
  Monitoring daily use of a speech generating device (SGD) for communication. Average communication rate based on total number of words used during the day.
Change in daily communication performance | 7 months vs. 8 months
  Monitoring daily use of a speech generating device (SGD) for communication. Average communication rate based on total number of words used during the day.
Change in daily communication performance | 8 months vs. 9 months
  Monitoring daily use of a speech generating device (SGD) for communication. Average communication rate based on total number of words used during the day.
Change in daily communication performance | 9 months vs. 10 months
  Monitoring daily use of a speech generating device (SGD) for communication. Average communication rate based on total number of words used during the day.
Change in daily communication performance | 10 months vs. 11 months
  Monitoring daily use of a speech generating device (SGD) for communication. Average communication rate based on total number of words used during the day.
Change in daily communication performance | 11 months vs. 12 months
  Monitoring daily use of a speech generating device (SGD) for communication. Average communication rate based on total number of words used during the day.
Change in daily communication performance | 12 months vs. 13 months
  Monitoring daily use of a speech generating device (SGD) for communication. Average communication rate based on total number of words used during the day.
Change in daily communication performance | 13 months vs. 14 months
  Monitoring daily use of a speech generating device (SGD) for communication. Average communication rate based on total number of words used during the day.
Change in daily communication performance | 14 months vs. 15 months
  Monitoring daily use of a speech generating device (SGD) for communication. Average communication rate based on total number of words used during the day.
Change in daily communication performance | 15 months vs. 16 months
  Monitoring daily use of a speech generating device (SGD) for communication. Average communication rate based on total number of words used during the day.
Change in daily communication performance | 16 months vs. 17 months
  Monitoring daily use of a speech generating device (SGD) for communication. Average communication rate based on total number of words used during the day.
Change in daily communication performance | 17 months vs. 18 months
  Monitoring daily use of a speech generating device (SGD) for communication. Average communication rate based on total number of words used during the day.
Change in daily communication performance | 18 months vs. 19 months
  Monitoring daily use of a speech generating device (SGD) for communication. Average communication rate based on total number of words used during the day.
Change in daily communication performance | 19 months vs. 20 months
  Monitoring daily use of a speech generating device (SGD) for communication. Average communication rate based on total number of words used during the day.
Change in daily communication performance | 20 months vs. 21 months
  Monitoring daily use of a speech generating device (SGD) for communication. Average communication rate based on total number of words used during the day.
Change in daily communication performance | 21 months vs. 22 months
  Monitoring daily use of a speech generating device (SGD) for communication. Average communication rate based on total number of words used during the day.
Change in daily communication performance | 22 months vs. 23 months
  Monitoring daily use of a speech generating device (SGD) for communication. Average communication rate based on total number of words used during the day.
Change in daily communication performance | 23 months vs. 24 months
  Monitoring daily use of a speech generating device (SGD) for communication. Average communication rate based on total number of words used during the day.

SECONDARY OUTCOMES:
User satisfaction of speech generating device (SGD) for daily communication | Baseline vs. 1 month
  Rating scale of user satisfaction with a range of 0-21 with a lower score representing a better outcome.
User satisfaction of speech generating device (SGD) for daily communication | 1 month vs. 2 months
  Rating scale of user satisfaction with a range of 0-21 with a lower score representing a better outcome.
User satisfaction of speech generating device (SGD) for daily communication | 2 months vs. 3 months
  Rating scale of user satisfaction with a range of 0-21 with a lower score representing a better outcome.
User satisfaction of speech generating device (SGD) for daily communication | 3 months vs. 4 months
  Rating scale of user satisfaction with a range of 0-21 with a lower score representing a better outcome.
User satisfaction of speech generating device (SGD) for daily communication | 4 months vs. 5 months
  Rating scale of user satisfaction with a range of 0-21 with a lower score representing a better outcome.
User satisfaction of speech generating device (SGD) for daily communication | 5 months vs. 6 months
  Rating scale of user satisfaction with a range of 0-21 with a lower score representing a better outcome.
User satisfaction of speech generating device (SGD) for daily communication | 6 months vs. 7 months
  Rating scale of user satisfaction with a range of 0-21 with a lower score representing a better outcome.
User satisfaction of speech generating device (SGD) for daily communication | 7 months vs. 8 months
  Rating scale of user satisfaction with a range of 0-21 with a lower score representing a better outcome.
User satisfaction of speech generating device (SGD) for daily communication | 8 months vs. 9 months
  Rating scale of user satisfaction with a range of 0-21 with a lower score representing a better outcome.
User satisfaction of speech generating device (SGD) for daily communication | 9 months vs. 10 months
  Rating scale of user satisfaction with a range of 0-21 with a lower score representing a better outcome.
User satisfaction of speech generating device (SGD) for daily communication | 10 months vs. 11 months
  Rating scale of user satisfaction with a range of 0-21 with a lower score representing a better outcome.
User satisfaction of speech generating device (SGD) for daily communication | 11 months vs. 12 months
  Rating scale of user satisfaction with a range of 0-21 with a lower score representing a better outcome.
User satisfaction of speech generating device (SGD) for daily communication | 12 months vs. 13 months
  Rating scale of user satisfaction with a range of 0-21 with a lower score representing a better outcome.
User satisfaction of speech generating device (SGD) for daily communication | 13 months vs. 14 months
  Rating scale of user satisfaction with a range of 0-21 with a lower score representing a better outcome.
User satisfaction of speech generating device (SGD) for daily communication | 14 months vs. 15 months
  Rating scale of user satisfaction with a range of 0-21 with a lower score representing a better outcome.
User satisfaction of speech generating device (SGD) or daily communication | 15 months vs. 16 months
  Rating scale of user satisfaction with a range of 0-21 with a lower score representing a better outcome.
User satisfaction of speech generating device (SGD) for daily communication | 16 months vs. 17 months
  Rating scale of user satisfaction with a range of 0-21 with a lower score representing a better outcome.
User satisfaction of speech generating device (SGD) for daily communication | 17 months vs. 18 months
  Rating scale of user satisfaction with a range of 0-21 with a lower score representing a better outcome.
User satisfaction of speech generating device (SGD) for daily communication | 18 months vs. 19 months
  Rating scale of user satisfaction with a range of 0-21 with a lower score representing a better outcome.
User satisfaction of speech generating device (SGD) for daily communication | 19 months vs. 20 months
  Rating scale of user satisfaction with a range of 0-21 with a lower score representing a better outcome.
User satisfaction of speech generating device (SGD) for daily communication | 20 months vs. 21 months
  Rating scale of user satisfaction with a range of 0-21 with a lower score representing a better outcome.
User satisfaction of speech generating device (SGD) for daily communication | 21 months vs. 22 months
  Rating scale of user satisfaction with a range of 0-21 with a lower score representing a better outcome.
User satisfaction of speech generating device (SGD) for daily communication | 22 months vs. 23 months
  Rating scale of user satisfaction with a range of 0-21 with a lower score representing a better outcome.
User satisfaction of speech generating device (SGD) for daily communication | 23 months vs. 24 months
  Rating scale of user satisfaction with a range of 0-21 with a lower score representing a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Katya Hill, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - AAC Institute Clinic (ICAN Talk Clinic), Carnegie, Pennsylvania
  - University of Pittsburgh, AAC Performance and Testing Laboratory, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee.